CLINICAL TRIAL: NCT02340520
Title: Enhancement of Corticosteroid Efficacy in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Nausherwan Burki, Professor of Medicine, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-032-3
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline; Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thophylline and roflumilast (Experimental): Theophylline for one week, followed by the addition of Roflumilast for a further one week.
  Interventions: Drug: Theophylline; Drug: Roflumilast

INTERVENTIONS:
Drug: Theophylline — Oral
Drug: Roflumilast — Oral

SUMMARY:
This is a pilot study designed to evaluate the effects of theophylline and roflumilast on circulating Histone deacetylase (HDAC) levels in subjects with COPD, and the bronchodilator effects of corticosteroids. Studies will be performed in 10 subjects with COPD nonresponsive to bronchodilators. Subjects will receive theophylline tablets for 1 week, followed by measurement of circulating HDAC and the acute effect of oral prednisone on the bronchodilator response to inhaled beta agonist. Roflumilast tablets will be added to the theophylline for a further week and the studies repeated. The study will provide preliminary data on the effects of theophylline and roflumilast on circulating HDAC levels and the effects of corticosteroids on the beta agonist bronchodilator response in COPD.

DETAILED DESCRIPTION:
1. SUBJECTS: 10 Stable patients >45 years of age, with an established diagnosis of COPD (18), with FEV1 <60% predicted, FEV1/FVC <70% and <+15% FEV1 response to bronchodilator will be recruited. Patients of both genders will be included.
2. TESTS

   a) Blood: i) HDAC 2 in peripheral blood mononuclear cells: ii) Serum theophylline level b) Spirometry for measurement of FVC, FEV1 and FEV1/FVC

   PROCEDURES Visit 1.
   1. After providing informed consent, subjects will receive a brief history and physical examination
   2. Blood will be drawn from a peripheral vein for HDAC2 levels (2 ml).
   3. Each subject will undergo baseline spirometry, which will be repeated after 3 inhalations of an albuterol inhaler.

   c) Subjects will be asked to continue their regular treatment regimen, including long and short acting beta agonists and anticholinergics, as well as inhaled steroids.

   d) Theophylline tablets extended-release 12 hr formulation, 300 mg orally taken every 12 hr will be dispensed, and the subject will return one week later for Visit 2. The subject will be asked to refrain from using his/her long acting beta agonists and anticholinergics for one day (24 hours) prior to Visit 2, and not to use the short acting beta agonist or take any caffeine containing drinks on the morning of visit 2. The subject will be asked to inform the P. I. should there be any adverse event.

   Subjects discontinuing the study drugs because of side effects will be withdrawn from the study.

   Visit 2.
   1. A brief history and physical examination will be performed and the subject will be asked about any change in symptoms.
   2. Blood (5 ml) will be drawn from a peripheral vein for HDAC2 and theophylline levels
   3. After baseline spirometry the subject will be given a single dose of 40 mg prednisone tablets.
   4. After 120 minutes, spirometry will be repeated, followed by 3 puffs of albuterol inhaler and repeat spirometry.

   The subject will then be asked to continue the theophylline tablets and in addition will be given roflumilast tablets 500 mcg orally once daily, and asked to return one week later for Visit 3.

   The subject will be asked to refrain from using his/her long acting beta agonists and anticholinergics for one day (24 hours) prior to Visit 3, and not to use the short acting beta agonist or take any caffeine containing drinks on the morning of visit 3. The subject will be asked to inform the P. I. should there be any adverse event.

   Visit 3
   1. A brief history and physical examination will be performed and the subject will be asked about any change in symptoms.
   2. Blood (5 ml) will be drawn from a peripheral vein for HDAC2 measurement.
   3. After baseline spirometry the subject will be given a single dose of prednisone tablets in a dose of 40 mg.
   4. After 120 minutes, spirometry will be repeated, followed by 3 puffs of albuterol inhaler and repeat spirometry.

   The subject will then have completed the study and will return to his/her previous treatment regimen.

   Data analysis:

   Results will be compared in terms of baseline vs drug by paired t test for change in FEV1 and FEV1/FVC as well as peripheral blood mononuclear blood HDAC2 levels. The relationship between FEV1 and FEV1/FVC and blood HDAC2 levels will be examined by correlation analysis.

   Expected results It is expected that with both theophylline and roflumilast treatment there will be a significant (p<0.05) increase in HDAC2 levels. It is also expected that with both theophylline and roflumilast treatment there will be a significant (p<0.05) increase in the bronchodilator response after the steroid dose, thereby supporting the hypothesis.

   It is also possible that there will be no effect on spirometry of either treatment; this would indicate that an increase in HDAC2 does not improve steroid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of COPD with FEV1 <60% predicted
* FEV1/FVC <70% and <+15% FEV1 response to bronchodilator.
* Patients of both genders will be included.
* IRB approved written informed consent will be obtained from each subject.

Exclusion Criteria:

1. Recent (<1 month) exacerbation of COPD,
2. Known hypersensitivity to beta agonists, theophylline, steroids, or roflumilast.
3. Current or recent (<2 weeks) treatment with oral steroids, theophylline or other methylxanthines, or roflumlast.
4. Diagnosis or history of asthma, uncontrolled hypertension, or congestive heart failure.
5. History of Cardiac arrhythmia
6. History of seizures.
7. History of Liver disease
8. Gastrointestinal disease, including history of peptic ulcer disease.
9. Current infection or antibiotic treatment.
10. History of depression or psychiatric disease.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nausherwan Burki, Principal Investigator — UConn Health
Locations (1):
- UConnHealth, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two of the 13 enrolled patients were found to be ineligible after being enrolled and therefore never started the study.
Groups:
- Theophylline and Roflumilast: Theophylline for one week, followed by the addition of Roflumilast for a further one week.
Period: Overall Study
Arm/Group | Theophylline and Roflumilast
Started | 11
Completed | 8
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Patient did not take drug as specified | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Three patients did not complete the study and therefore their data was removed from the analyses.
Arm/Group | Theophylline and Roflumilast
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic/Latino | 7
  African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Bronchodilation
Description: Change in FEV1 L and FVC L
Time Frame: Baseline, Week 1 and 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Theophylline and Roflumilast
Number analyzed (Participants) | 8
liters
  baseline FEV1 | 1.18 (0.51)
  baseline FVC | 2.72 (0.78)
  week 1 FEV1 | 1.22 (0.51)
  week 1 FVC | 2.90 (0.82)
  post steroid week 1 FEV1 | 1.18 (0.51)
  post steroid week 1 FVC | 2.72 (0.68)
  week 2 FEV1 | 1.25 (0.58)
  week 2 FVC | 2.79 (0.71)
  week 2 post steroid FEV1 | 1.18 (0.51)
  week 2 post steroid FVC | 2.81 (0.61)
  week 1, FEV1 post bronchodilator, post steroid | 1.24 (0.54)
  week 1, FVC post bronchodilator, post steroid | 2.80 (0.65)
  week 2, FEV1 post bronchodilator, post steroid | 1.30 (0.47)
  week 2, FVC post bronchodilator, post steroid | 2.98 (0.67)
Statistical Analysis 1: Comparison: Theophylline and Roflumilast; Test type: Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Change in HDAC2 Levels
Description: circulating Histone Deacetylase2 levels measured in blood sample
Time Frame: Baseline, Week 1 and 2
Measure: Mean (Standard Error); unit: µM/µg
Arm/Group | Theophylline and Roflumilast
Number analyzed (Participants) | 8
µM/µg
  baseline | 2.96 (0.73)
  week 1 | 2.58 (0.91)
  week 2 | 2.81 (0.40)
Statistical Analysis 1: Comparison: Theophylline and Roflumilast; Test type: Other; p > 0.1, ANOVA

ADVERSE EVENTS:
Arm/Group | Theophylline and Roflumilast
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No